CLINICAL TRIAL: NCT02357381
Title: eNeura SpringTMS Post-Market Observational U.S. Study of Migraine
Brief Title: eNeura SpringTMS Post-Market Observational US Study of Migraine
Acronym: ESPOUSE
Status: Completed | Type: Observational
Sponsor: eNeura, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SpringTMSUSPMOS 2014-01
Record Dates: First submitted 2015-02-03; First posted 2015-02-06 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2015-04

CONDITIONS: Headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- TMS Treatment: TMS( transcranial magnetic stimulation) -treatment for headache
  Interventions: Device: eNeura SpringTMS

INTERVENTIONS:
Device: eNeura SpringTMS — Single pulse magnetic stimulation for prevention and/or treatment of migraine headache with or without aura.

SUMMARY:
A multi-center, prospective, non-randomized, single arm, open label, post-market, observational study to evaluate the use of the eneura, springtms system in reduction of migraine headache symptoms.

DETAILED DESCRIPTION:
A prospective, non-randomized, single arm, multi-center observational study designed to evaluate the use of the SpringTMS system in reducing the frequency of headache days.

Note: This is a NON-SIGNIFICANT RISK (NSR) study of a NON-SIGNIFICANT RISK (NSR) Device. It is a post market study of a NSR device cleared by FDA through the 510(k) pre-market notification process. The cleared indications for use are provided above. This NSR study is designed to collect information on additional applications of the SpringTMS device. These additional applications include:

1. Use of the device to evaluate the potential for regular use of sTMS to reduce the frequency, severity, and/or duration of migraine.
2. Delivery of additional treatments (pulses) to evaluate the acute treatment efficacy of breakthrough migraine attacks with and without aura.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 to 65 years of age;
2. Patients able to understand and communicate in English;
3. Migraine with or without aura;
4. 4-25 headache days per month (confirmed by 1-month baseline diary, minimum of 5 complete headache-free days/month);
5. Understand and willing to provide diary and survey data.

Exclusion Criteria:

* Subjects will be excluded from participating in this trial if they meet any of the following criteria

  1. Severe co-existing disease having a life expectancy of less than 1 year;
  2. Currently involved in any other investigational clinical trials that have not completed their primary endpoint or that may interfere with the SpringTMS study results;
  3. Mental impairment or other conditions which may not allow the subject to understand the nature, significance and scope of the study and to cooperate with follow-up requirements;
  4. Known drug and/or alcohol addiction or use of illicit substances;
  5. Patients with epilepsy or history of seizure;
  6. Severe active major depression or major psychiatric illness;
  7. Concurrent use of other neurostimulation devices (Cefaly®, TENS, implantable devices);
  8. Use of Botox® within past 4 months;
  9. Extracranial nerve block (e.g. occipital, supraorbital) within past 3 months;
  10. Use of Cefaly for prevention within past month;
  11. Patients with metal containing implants as follows:

The SpringTMS may not be used in patients who have metals, conductive materials, or metal-containing implants in their head, neck or upper body. Patients with implants that are affected by a magnetic field should not use the SpringTMS. Examples of such implants include:

* Aneurysm clips or coils • Radioactive seeds
* Cochlear implants • Magnetically programmable shunt valves
* Cerebral spinal fluid shunts • Stents
* Bullets or pellets lodged in the head or upper body • Metal plates, screws, staples or sutures in skull, neck, shoulders, arms or hands
* Filters • Metallic artificial heart valves
* Electrodes • Facial tattoos with metallic ink Dental implants, fillings, or other dental appliances are okay and are not affected by the device.

Note: although not explicitly excluded, safety and effectiveness have not been established in pregnant women. Please defer to the judgment of the investigator when considering the eligibility of this population.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 4-25 headache days per month (confirmed by 1-month baseline diary, minimum of 5 complete headache-free days/month)
Sampling Method: Non-Probability Sample
Enrollment: 263 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2016-07-01 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Headache Days | 3 months
  Reduction in mean headache days

CONTACTS AND LOCATIONS:
Overall Officials: David W Dodick, MD, Principal Investigator — Mayo Clinic , Phoenix,AZ
Locations (7):
- United States (7):
  - Mayo Clinic, Phoenix, Arizona
  - UCLA Headache Research and Treatment Program, Los Angeles, California
  - Stanford Headache Program, Stanford, California
  - Mid Atlantic Permanente Medical Group-Kaiser, Rockville, Maryland
  - Albert Einstein College of Medicine, The Bronx, New York
  - The Cleveland Clinic Center for Headache and Pain, Cleveland, Ohio
  - Jefferson Headache Center, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Starling AJ, Tepper SJ, Marmura MJ, Shamim EA, Robbins MS, Hindiyeh N, Charles AC, Goadsby PJ, Lipton RB, Silberstein SD, Gelfand AA, Chiacchierini RP, Dodick DW. A multicenter, prospective, single arm, open label, observational study of sTMS for migraine prevention (ESPOUSE Study). Cephalalgia. 2018 May;38(6):1038-1048. doi: 10.1177/0333102418762525. Epub 2018 Mar 4. PMID 29504483